CLINICAL TRIAL: NCT03909672
Title: Cupping Therapy in the Treatment of Individuals With Nonspecific Chronic Low Back Pain
Brief Title: Cupping Therapy in Nonspecific Chronic Low Back Pain
Acronym: cupping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Marcelo Cardoso de Souza, PT, PhD., Professor, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UFRNventosa
Record Dates: First submitted 2019-04-06; First posted 2019-04-10 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Low Back Pain
Keywords: low back pain; cupping therapy
MeSH Terms: conditions — Low Back Pain | interventions — Cupping Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cupping therapy with 2 suctions (Experimental): Participants in the intervention group will receive the application of cupping therapy with two acrylic type 1 cups with a distance of 3 cm each cup, parallel to the L1 to L5 vertebrae bilaterally. This group will consist of the application of windsheets with 2 suctions for 10 minutes, once a week, for 10 weeks. The cups shall be secured by means of elastic bands.
  Interventions: Other: Cupping Therapy
- Cupping Therapy sham (Placebo Comparator): The placebo group will receive the application of cupping therapy with 2 cups of acrylic type size 1 with a distance of 3 cm each cup, parallel to the vertebrae L1 to L5, bilaterally . This group will consist of applying the sham winds for 10 minutes, once a week for 10 weeks.
  However, the cups will be made with small holes <2 mm in diameter to release the negative pressure in seconds. The cups will also be fixed by means of elastic bands.
  Interventions: Other: Cupping Therapy

INTERVENTIONS:
Other: Cupping Therapy — application of cupping therapy with two acrylic type 1 cups (4.5 cm internal diameter, Dong Yang ® brand) with a distance of 3 cm each cup, parallel to the L1 to L5 vertebrae bilaterally

SUMMARY:
Introduction: Low back pain is a very prevalent condition in the population and windsurf therapy has been presented as a non-pharmacological treatment currently used in this population. However, there is a lack of studies that evaluate such effects, besides a standardization of application of the technique in this condition. This protocol describes a placebo-controlled, randomized, double-blind study that aims to assess the effectiveness of windsurf therapy in improving pain and other symptoms of individuals with chronic non-specific back pain. Methods: Ninety individuals with chronic nonspecific and localized chronic low back pain from 18 to 59 years, will be recruited according to the inclusion criteria. Afterwards they will be randomized to one of the 2 groups: intervention group (GI) where it will be submitted applied to the windspiration with 2 suctions; and placebo group (GP) with simulated application. Both applications will occur in parallel to the vertebrae from L1 to L5 bilaterally. The application will be performed once a week for eight weeks. The volunteers will be evaluated before treatment (T0), immediately after the first intervention (T1), 4 weeks after treatment (T4) and 8 weeks after treatment (T8). The primary endpoint will be pain, and the secondary ones will be kinesiophobia, physical function, lumbar range of motion, sleep quality, patient expectation, quality of life, and psychological factors. Discussion: This is the first protocol that proposes to evaluate the effect of windsotherapy on lumbar ROM, sleep quality, kinesiophobia and psychological problems. Few studies have been done on windsurfing individuals with low back pain, requiring further studies with good methodological quality. Because there is no consensus on the use of windsurf therapy in individuals with nonspecific chronic low back pain, our protocol will be the basis for the use of the technique by health professionals and for new studies to be performed.

DETAILED DESCRIPTION:
This study will involve 4 researchers; 1 researcher responsible for evaluations; 1 researcher responsible for interventions; 1 researcher responsible for the interview, initial screening and randomization of participants, and 1 researcher who will perform the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* female and male individuals aged between 18 and 59 years, normal BMI, presenting localized and non-specific lower back pain for more than 3 months;
* have not used cupping therapy before;
* report pain between 3 and 8 by NRS;
* individuals who are not under physiotherapeutic treatment during the intervention;
* individuals without neurological, vestibular, visual or auditory deficits that make evaluations impossible.

Exclusion Criteria:

* Individuals with cutaneous lesions in the region where they will be applied to cupping therapy,
* Individuals with uncontrolled diabetes and hypertension;
* Irradiated and sacral lumbar pain;
* Individuals with contraindication to windsurf therapy, are: cancer, renal failure, hepatic and cardiac insufficiency, pacemaker, pregnancy;
* Individuals with severe spinal pathology (including fractures, inflammatory diseases and tumors);
* Travel planning in the next 2 months

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Change from Numeric Rating Scale (NRS) of Pain | T0 -baseline, T4 (four week) and T8 (eight week)
  The patients are asked to circle the number between 0 and 10. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'

SECONDARY OUTCOMES:
Change from Oswestry Disability Index (ODI) | T0 -baseline and T8 (eight week)
  will be used to analyze the quality of life in people with low back pain. This instrument contains in 10 items that assess the impact of low back pain on several functional activities. Values range from 0 to 5, the highest value indicating greater disability. The end result is the sum of all items.
Range of motion of the lower back (ROM) | T0 -baseline, T4 (four week) and T8 (eight week)
  Will be evaluated through the finger-to-floor test. This test presents high reliability and can be used for clinical practice and scientific studies.
Short-Form 36 questionnaire (SF-36) | T0 -baseline and T8 (eight week)
  Quality of life will be assessed by the Short-Form 36 (SF-36) questionnaire. The instrument consists of 36 questions and assesses eight different domains that influence quality of life, considering the individual's perception of their health aspects in the last four weeks. Each item has a group of answers distributed on a Likert-graded scale, and the following dimensions were evaluated: physical function, physical aspect, pain, general health, vitality, social function, emotional aspect and mental health. Your total score ranges from 0 to 100, where the higher the value, the better quality of life score.
Timed Up and Go Test (TUG): | T0 -baseline and T8 (eight week)
  This is a functional test which quantifies the mobility of an individual in seconds through the time in which they perform the task, i.e. in how many seconds can they lift themselves from a chair, walk 3 meters, turn, return to the chair, and sit down again. The test has already been used in individuals to assess function in individuals with low back pain. The shorter the time taken to perform a task, the better the individual's ability to perform.
Global Perceived Effect Scale (GPE) | T8 (eight week)
  Is a direct scale about the patient's self-perception when the intervention is performed.The GPE evaluates using 11 points, starting from a negative 5 (much worse than when starting the treatment), a neutral rating of 0, and 5 is positive (much improvement from starting the treatment). The Portuguese version will be used. The GPE evaluates using 11 points, starting from a negative 5 (much worse than when starting the treatment), a neutral rating of 0, and 5 is positive (much improvement from starting the treatment) .
Hospital Anxiety and Depression Scale (HADS) | T0 -baseline and T8 (eight week)
  A questionnaire which has also been validated and translated into Portuguese. This scale has 14 items, 7 for anxiety subscale and 7 for depression. For each item there is a score of 0 to 3, with a total of 21 points for the scale.
Medication consumption | T8 (eight week)
  Patients will be given a daily control list of medication use to mark the amount of their use for low back pain during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Cardoso De Souza, PT,PhD, Study Chair — Universidade Federal do Rio Grande do Norte
Locations (1):
- Marcelo Souza, Santa Cruz, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No
there isn't a plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Wang YT, Qi Y, Tang FY, Li FM, Li QH, Xu CP, Xie GP, Sun HT. The effect of cupping therapy for low back pain: A meta-analysis based on existing randomized controlled trials. J Back Musculoskelet Rehabil. 2017 Nov 6;30(6):1187-1195. doi: 10.3233/BMR-169736. PMID 28946531
- [Result] Moura CC, Chaves ECL, Cardoso ACLR, Nogueira DA, Correa HP, Chianca TCM. Cupping therapy and chronic back pain: systematic review and meta-analysis. Rev Lat Am Enfermagem. 2018 Nov 14;26:e3094. doi: 10.1590/1518-8345.2888.3094. PMID 30462793
- [Derived] Almeida Silva HJ, Barbosa GM, Scattone Silva R, Saragiotto BT, Oliveira JMP, Pinheiro YT, Lins CAA, de Souza MC. Dry cupping therapy is not superior to sham cupping to improve clinical outcomes in people with non-specific chronic low back pain: a randomised trial. J Physiother. 2021 Apr;67(2):132-139. doi: 10.1016/j.jphys.2021.02.013. Epub 2021 Mar 20. PMID 33757719
- [Derived] Silva HJA, Saragiotto BT, Silva RS, Lins CAA, de Souza MC. Dry cupping in the treatment of individuals with non-specific chronic low back pain: a protocol for a placebo-controlled, randomised, double-blind study. BMJ Open. 2019 Dec 22;9(12):e032416. doi: 10.1136/bmjopen-2019-032416. PMID 31871257
- Available data/document: Study Protocol — http://facisa.ufrn.br